CLINICAL TRIAL: NCT03688802
Title: A Single-Center, Randomized, Controlled, Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Goblet Cell and Meibomian Gland Stimulation (The IMPERIAL Study)
Brief Title: Efficacy of OC-01 Nasal Spray on Goblet Cell and Meibomian Gland Stimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-005
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OC-01 (varenicline) nasal spray, 1.2 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 1.2 mg/mL, one time dosing
  Interventions: Drug: OC-01 (varenicline) nasal spray
- Placebo (vehicle control) nasal spray (Placebo Comparator): Placebo (vehicle control) nasal spray, one time dosing
  Interventions: Drug: Placebo (vehicle control) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline) nasal spray — OC-01 (varenicline) nasal spray
  Arms: OC-01 (varenicline) nasal spray, 1.2 mg/mL
Drug: Placebo (vehicle control) nasal spray — Placebo
  Arms: Placebo (vehicle control) nasal spray

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-01 Nasal Spray as compared to placebo in simulating Goblet Cell and Meibomian Gland function in adult subjects with DED.

DETAILED DESCRIPTION:
This was a Phase 2, single-center, randomized, masked (including all subjects, investigators, and study site personnel), placebo-controlled study designed to evaluate the safety and efficacy of OC-01 (varenicline) nasal spray in stimulating goblet cell and Meibomian gland function in in adult subjects with DED. Approximately 45 subjects at least 18 years of age with a physicians' diagnosis of DED and meeting all other study eligibility criteria were planned to be randomized to receive a single application of 0.2% (1.2 mg/mL) OC-01 or placebo

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to visit 1.

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery (e.g. laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dieckmann GM, Cox SM, Lopez MJ, Ozmen MC, Yavuz Saricay L, Bayrakutar BN, Binotti WW, Henry E, Nau J, Hamrah P. A Single Administration of OC-01 (Varenicline Solution) Nasal Spray Induces Short-Term Alterations in Conjunctival Goblet Cells in Patients with Dry Eye Disease. Ophthalmol Ther. 2022 Aug;11(4):1551-1561. doi: 10.1007/s40123-022-00530-x. Epub 2022 Jun 2. PMID 35653029

RESULTS

PARTICIPANT FLOW:
Groups:
- OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL: OC-01 (varenicline) nasal spray, 1.2 mg/mL
  OC-01 (varenicline) nasal spray: OC-01 (varenicline) nasal spray
- Placebo (Vehicle Control) Nasal Spray: Placebo (vehicle control) nasal spray
  Placebo (vehicle control) nasal spray: Placebo
Period: Overall Study
Arm/Group | OC-01 (Varenicline) Nasal Spray, 1.2 mg/mL | Placebo (Vehicle Control) Nasal Spray
Started | 12 | 6
Completed | 11 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OC-01, 1.2 mg/mL: OC-01: OC-01 (varenicline) nasal spray
- Placebo: Placebo (vehicle) nasal spray: Placebo
- Total: Total of all reporting groups
Arm/Group | OC-01, 1.2 mg/mL | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (13.79) | 63.3 (13.46) | 61.4 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 6 | 17
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18
Schirmer's Test Score [Mean (Standard Deviation); unit: mm] — Schirmer's Test Score from 0-35 mm where a higher score is indicative of a better outcome.
  mm | 6.6 (4.42) | 4.5 (3.89) | 5.9 (4.25)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Goblet Cell Area
Description: Mean change in Goblet Cell Area with a larger decrease is indicative of a better outcome.
Time Frame: Baseline (pre-treatment), 1 day (post treatment)
Population: Subjects in the ITT population. Only Subjects who had both pre-treatment and post-treatment values were utilized in the change from pre-treatment statistics.
Measure: Mean (Standard Deviation); unit: um
Groups:
- Placebo: Placebo: Placebo Vehicle ) nasal spray
Arm/Group | OC-01, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 7 | 3
um | -38.8 (30.20) | -6.7 (1.94)

2. Primary Outcome: Mean Change in Goblet Cell Perimeter
Description: Mean change in Goblet Cell Perimeter. A larger decrease is indicative of a better outcome.
Time Frame: Baseline (pre-treatment), 1 day (post treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: um
Arm/Group | OC-01, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 7 | 3
um | -7.7 (5.79) | -1.8 (0.76)

3. Primary Outcome: Change in Meibomian Gland Area, Upper Lid
Description: Change in Meibomian gland area, upper lid. A larger decrease is indicative of a better outcome
Time Frame: Baseline (pre-treatment), 1 day (post treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: um
Arm/Group | OC-01, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 10 | 6
um | 11.2 (118.6) | -143.2 (154.8)

4. Primary Outcome: Mean Change in Meibomian Gland Area, Lower Lid.
Description: Mean change in Meibomian Gland Area, lower Lid. A larger decrease is indicative of a better outcome.
Time Frame: Baseline (pre-treatment), 1 day (post treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: um
Arm/Group | OC-01, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 9 | 6
um | -29.9 (88.1) | -12.4 (95.8)

5. Primary Outcome: Mean Change in Meibomian Gland Perimeter, Upper Lid.
Description: Chane in Meibomian Gland Perimeter, upper lid. A larger decrease is indicative of a better outcome.
Time Frame: Baseline (pre-treatment), 1 day (post treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: um
Arm/Group | OC-01, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 10 | 6
um | 6.15 (16.6) | -19.2 (22.8)

6. Primary Outcome: Mean Change in Meibomian Gland Perimeter, Lower Lid
Description: Mean change in Meibomian Gland Perimeter, lower lid. A larger decrease is indicative of a better outcome.
Time Frame: Baseline (pre-treatment), 1 day (post treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: um
Arm/Group | OC-01, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 9 | 6
um | -4 (10.9) | 4.2 (19.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration to the last study visit (pre to post treatment 1 day).
Groups:
- OC-01, 1.2 mg/mL: OC-01 (varenicline) nasal spray, 1.2 mg/mL
- Placebo: Placebo (vehicle control) nasal spray
Arm/Group | OC-01, 1.2 mg/mL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 6/12 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC-01, 1.2 mg/mL (N=12) | Placebo (N=6)
TEAE (Eye disorders) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03688802/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03688802/SAP_002.pdf